CLINICAL TRIAL: NCT01391390
Title: The Effect of Melatonin Treatment on Tardive Dyskinesia and Oxidative Stress: A Double-Blind Placebo-Controlled Trial
Brief Title: Melatonin Treatment for Tardive Dyskinesia in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing HuiLongGuan Hospital (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Xiang Yang Zhang, Director, Biological Psychiatry Center, Beijing HuiLongGuan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BJ-7072035
Record Dates: First submitted 2011-07-07; First posted 2011-07-12 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Tardive Dyskinesia
Keywords: Tardive Dyskinesia; Schizophrenia; Melatonin; Oxidative Stress; Antioxidant
MeSH Terms: conditions — Tardive Dyskinesia; Schizophrenia | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Melatonin, antioxidant, oxidative stress (Experimental): Melatonin is an active treatment for TD.
  Interventions: Drug: Melatonin
- Placebo (Placebo Comparator): Placebo look like the active drug, and same dose.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Melatonin — 10mg/day, 12-week treatment
  Other Names: APRD00742
  Arms: Melatonin, antioxidant, oxidative stress
Drug: Placebo — 10mg/day, 12-week treatment for TD
  Arms: Placebo

SUMMARY:
This is a double-blind, randomized, placebo-controlled trial of melatonin as an add-on therapy to antipsychotics will be performed to examine the effects of melatonin on tardive dyskinesia symptoms and cognitive deficits in 120 patients with established tardive dyskinesia (TD). This study addresses a free radical hypothesis of TD.

DETAILED DESCRIPTION:
1. Since it has been proposed that neuroleptic-induced increases in free-radical production may relate to the development of TD, the investigators hypothesize that melatonin, an effective antioxidant, may attenuate the severity of tardive dyskinesia symptoms.
2. Due to increased cognitive deficits in patients with TD and implication of oxidative stress in cognitive impairment, the investigators hypothesize that both cognitive impairment and tardive dyskinesia symptoms may be induced by the same pathophysiological stimulus--oxidative stress. Hence, the investigators further hypothesize that both tardive dyskinesia symptoms and cognitive deficits in patients with TD may be improved by melatonin simultaneously.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of both schizophrenia and TD;
2. duration of TD symptoms longer than 1 year;
3. on stable doses of antipsychotic drug for at least 6 months;
4. between 18 and 70 years of age.

Exclusion Criteria:

1. comorbid neurological illness other than TD;
2. if they have received vitamin C or vitamin E within 1 month before the start of the study;
3. alcohol/drug abuse;
4. acute, unstable medical condition;
5. pregnant or breastfeeding female;
6. use of other antioxidants.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-09; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
the Abnormal Involuntary Movement Scale (AIMS) | 12 weeks

SECONDARY OUTCOMES:
the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | 12 weeks
the Positive and Negative Syndrome Scale (PANSS) | 12 weeks
the Simpson-Angus Scale for extrapyramidal side effects (SAS) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lian Y Cao, MD, Study Chair — Beijing HuiLongGuan Hospital
Locations (1):
- Beijing HuiLongGuan hospital, Beijing, China